CLINICAL TRIAL: NCT06883175
Title: Evolution of the Chicago Classification: Bridging Physiology and Mechanics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: The California Medical Innovations Institute, Inc. (Other)
Responsible Party: Principal Investigator, John Pandolfino, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCv5
Record Dates: First submitted 2024-11-25; First posted 2025-03-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dysphagia; Achalasia, Esophageal; Ineffective Esophageal Motility
Keywords: dysphagia; swallowing
MeSH Terms: conditions — Deglutition Disorders; Esophageal Achalasia | interventions — prucalopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dysphagia participants (Experimental): There are no arms in this study. All subjects will be studied in like manner.
  Interventions: Diagnostic Test: FLIP; Diagnostic Test: HRM; Other: Prucalopride

INTERVENTIONS:
Diagnostic Test: FLIP — Functional Lumen Impedance Planimetry
Diagnostic Test: HRM — HIgh Resolution Manometry
Other: Prucalopride — Medication

SUMMARY:
Swallowing difficulties are extremely common and result in substantial morbidity, reduction in the quality of life, and mortality related to malnutrition and complications from regurgitation and aspiration. Unfortunately, our understanding regarding the pathophysiology of dysphagia and GERD has been hampered by focusing predominantly on circular muscle activity and ignoring the essential biomechanical properties of the esophageal wall that promote normal emptying. Our initial work explored the relationship between intrabolus pressure (IBP) and esophagogastric junction (EGJ) compliance as a metric for outflow resistance. This work highlighted the direct relationship between IBP and EGJ opening and was the foundation for the development of the classification scheme utilized around the world to diagnose esophageal motor disorders: "the Chicago Classification" (CC). Despite this improved understanding focused on bolus transit dynamics, there are still significant gaps in our scientific understanding centered on the lack of a true correlate for symptoms, reliable predictive models and effective treatments for Functional dysphagia, IEM and EGJOO. Given these limitations, we have developed novel approaches that combine assessments of primary and secondary peristalsis (a NeuroMyogenic Model of esophageal function). These will leverage our recent findings supporting the importance of the esophageal response to distension in bolus clearance, noting that this response of the esophageal wall to bolus retention or reflux is one of the most essential functions of the esophagus in preventing complications of aspiration, or reflux injury. We will also include an assessment of esophageal geometry and wall biomechanics (elasticity/dilatation) as these carry essential interactions with esophageal function that are overlooked in the current diagnostic paradigms.

In order to test our hypothesis that wall mechanics are a major determinant of esophageal diseases, we had to develop new approaches and new technology to directly measure mechanical wall state, descending inhibition and LES opening. Using impedance techniques combined with manometry, we are now capable of assessing IBP and diameter changes across a space-time continuum (4D HRM). We also developed physics-based hybrid diagnostics that include a FLIP technique to assess esophageal work and power during volumetric distention (FLIP-MECH) and a fluoroscopy approach that simultaneously assesses esophageal diameter-pressure relationships (Fluoro-MECH). We also developed a new approach, Interactive FLIP Panometry, which facilitates an assessment of descending inhibition and the mechanism behind impaired LES opening. These tools will allow us to expand our models to combine an assessment of neuromyogenic function simultaneously with geometry. Our overarching goal will be to study well-defined patient populations (Functional Dysphagia, IEM/GERD, EGJOO and Achalasia) before and after targeted interventions to test the NeuroMyogenic and MechanoGeometric Model. This work will build upon the previous success of the CC and help advance the evolution of the CC by defining new, relevant biomechanical physiomarkers of disease activity that can identify new targets for therapeutic intervention and facilitate prediction of clinical outcomes.

DETAILED DESCRIPTION:
The proposed experiments in this application will utilize both standard of care diagnostic testing and treatment as well as research procedures in small subsets of participants as required for each Specific Aim. No randomization will be utilized in any aim. The source of the study population will be male and female subjects aged 18-85 years old inclusive and mentally capable to provide informed consent who present to the Northwestern Medicine Digestive Health Center with the chief complaint of dysphagia, regurgitation, chest pain or food impaction, or referral for treatment of achalasia, GERD, or endoscopy negative dysphagia. These subjects will be approached by the study team and provide informed consent prior to study involvement.

In Aim 1, 375 subjects (300 with FD, IEM, or EGJOO and 75 with GERD) will participate. For Aim 1a, standard of care procedural results and questionnaires will be used to develop the best thresholds that will stage the NeuroMyogenic Model. Sixty of these subjects will undergo open-label treatment with prucalopride (2mg qD (oral) for 2 weeks) with completion of questionnaires (research) after the 2 week time period. Fifteen of these (5 each stage of the Neuromyogenic model- I, II, and III) will complete a post-treatment procedure visit where they will undergo sedated FLIP with manometry and esophagram evaluation with questionnaires on the last day of medication. Sample sizes for this experiment are based on our previous results, where patients with HRM of normal motility, IEM, or AC will yield NeuroMyogenic classification of stage I in 15%, stage II in 15%, and stage III in 10% (with 60% of patients being "normal function dysphagia"), thus sample sizes of n=20 for each group will be feasible for recruitment.

For Aim 1b, we will recruit 50 subjects with IEM/FD with impaired LES Opening on FLIP and 50 with EGJOO and assess the ability of EUS-guided Botox to relieve symptoms as measured by EGJ opening before and after treatment. Additionally, a comparison group of type II achalasia (n=15) without significant dilatation (esophageal width <3cm) will be tested with Interactive FLIP Panometry (Comparison from Aim 2a). Based on our data, we anticipate 20% of 250 patients with HRM of normal motility, IEM, or AC will have abnormal EGJ opening. The response rate to distension and botulinum toxin are not a priori known for EGJOO or FD patients, thus, considering rates from 15-90%, our planned sample size of n=50 per group would provide 80% power to detect absolute differences between groups of 13-27%, which correspond to odds ratios of 3.0-6.9.

For Aim 1c, 75 subjects with GERD will undergo pH-impedance testing, HRM, FLIP and complete PROs as part of their standard of care before and after treatment (fundoplication or MSA). HRM is performed prior to the placement of the pH-Impedance catheter and the HRM procedural data along with FLIP data will be used in this experiment to attempt to predict the likelihood of dysphagia (as measured by BEDQ) after MSA or fundoplication. Assuming 25-50% of patients develop dysphagia and abnormal bolus transit occurs in 13-31% of these patients, our model would have 80% power to detect effects on the order of odds ratios of 2.6-3.3.

Aim 2 experiments focus on achalasia as the disease of interest and explore the role of abnormal geometry and esophageal wall state in determining clinical outcomes of treatment and esophageal emptying. Subjects will be studied using our clinical physiomechanical protocol (EGD, FLIP, HRM, TBE) as part of their standard of care before and 6 months after short tailored POEM. Two hundred subjects will be studied. The primary outcomes will be esophageal clearance and recoil (elasticity) in 100 subjects for experiment 2a. These data will be subject to a supervised learning method to define thresholds for defining the stages of achalasia. The planned cohort sizes (n=100) have traditionally been sufficient for fitting and evaluating SVM.

In experiment 2b, the SOC information will be collected from all 200 subjects and used to measure the primary outcome of treatment success defined as Eckart Score <3 and TBE 5-min column height <5cm (without re-intervention). We will study the success of POEM when the EGJ-Distensibility threshold is set at 3.0. Patients who fail will undergo repeat POEM to a target EGJ-DI of 6.0. We theorize that the higher stages will require a higher target for EGJ-DI. Assuming up to 10% attrition, GLM using all n=200 patients would have 80% power to detect differences in treatment response rates across up to 5 stages consistent with those rates ranging from 60-90%.

ELIGIBILITY:
Inclusion Criteria:

* The source of the study population will be male and female subjects aged 18-85 years old inclusive (females of childbearing potential should be on highly effective contraceptive methods) and mentally capable to provide informed consent who present to the Northwestern Medicine Digestive Health Center with the chief complaint of dysphagia, regurgitation, chest pain or food impaction, or referral for treatment of achalasia, GERD, scleroderma, or endoscopy negative dysphagia. All subjects must be able to undergo endoscopy with functional lumen imaging probe (FLIP) and transnasal intubation for 4 dimensional-High Resolution Manometry (4D HRM) and 24-hour pH impedance probe.

Exclusion Criteria:

* Currently participating in a concurrent clinical trial or completed another trial within past 8 weeks.

  * Active severe esophagitis (Los Angeles esophagitis Grade C and above), Patients may be eligible once esophagitis is healed if they continue to have dysphagia in the context of healed esophagitis.

Contact PD/PI: Pandolfino, John Erik Protection of Human Subjects Page 131

* Evidence of mechanical obstruction due to stricture (e.g., peptic/GERD patients, EoE, or other) or previous small bowel or colonic obstruction.
* Long-segment Barrett's metaplasia.
* Unstable medical illness with ongoing diagnostic work-up and treatment. Patients with well-controlled hypertension, diabetes and a remote history of ischemic heart disease that is deemed stable, as judged by the physician-investigator can be included. EKG will be performed before prucalopride in the 60 patients undergoing Experiment 1a.
* Current drug or alcohol abuse or dependency.
* Current neurologic or cognitive impairment which would make the patient an unsuitable candidate for a research trial.
* Severe mental illness, e.g., uncontrolled major depression with suicidal ideation, active psychosis, diagnosis of schizophrenia-spectrum disorder.
* Pregnant patients.
* Bleeding diathesis or need for anticoagulation that cannot be stopped for endoscopy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Brief Esophageal Dysphagia Questionnaire (BEDQ) | baseline
  A 10 item dysphagia/food impaction questionnaire measured on a 6-point Likert scale from "none" to "severe" with higher scores indicating a greater degree of dysphagia
Brief Esophageal Dysphagia Questionnaire (BEDQ) | 6 months post-treatment
  A 10 item dysphagia/food impaction questionnaire measured on a 6-point Likert scale from "none" to "severe" with higher scores indicating a greater degree of dysphagia
Esophagogastric Junction (EGJ) diameter | baseline
  Measurement of EGJ diameter in cm
Esophagogastric Junction (EGJ) diameter | 6 months post-treatment
  Measurement of EGJ diameter in cm
Esophageal Clearance | baseline
  Barium column height of 0 cm at 5 minutes
Esophageal Clearance | 6 months post-treatment
  Barium column height of 0 cm at 5 minutes
recoil | baseline
  decrease in wall diameter >1cm
recoil | 6 months post-treatment
  decrease in wall diameter >1cm
Timed Barium Esophagram (TBE) Column Height | baseline
  Height of barium column at 5 minutes (Timed Barium Esophagram)
Timed Barium Esophagram (TBE) Column Height | 6 months post-treatment
  Height of barium column at 5 minutes (Timed Barium Esophagram)
Integrated Relaxation Pressure (IRP) | baseline
  Mean EGJ pressure for 4 seconds of relaxation in the ten-second window following deglutitive Upper Esophageal Sphincter relaxation relaxation.
Integrated Relaxation Pressure (IRP) | 6 months post-treatment
  Mean EGJ pressure for 4 seconds of relaxation in the ten-second window following deglutitive Upper Esophageal Sphincter relaxation
Esophagogastric Junction Distensibility Index | baseline
  A measure of the distensibility of the EGJ using Functional Luminal Impedance Probe
Esophagogastric Junction Distensibility Index | 6 months post-treatment
  A measure of the distensibility of the EGJ using Functional Luminal Impedance Probe

SECONDARY OUTCOMES:
Bolus Retention | baseline
  A combined measurement of barium column height (in cm) at 5 minutes (Timed Barium Esophagram) and Impedance Bolus Height (4D HRM)
Bolus Retention | 6 months post-treatment
  A combined measurement of barium column height (in cm) at 5 minutes (Timed Barium Esophagram) and Impedance Bolus Height (4D HRM)
Eckhart Score | baseline
  A 4-item self-report scale measuring weight loss, chest pain, regurgitation, and Dysphagia. Scores range 0-4, lower is better.
  chest pain, regurgitation, and dysphagia
Eckhart Score | 6 months post-treatment
  A 4-item self-report scale measuring weight loss, chest pain, regurgitation, and Dysphagia. Scores range 0-4, lower is better.
  chest pain, regurgitation, and dysphagia

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdi H, Williams LJ. Principal component analysis. WIREs Computational Statistics. 2010;2(4):433-59. doi: 10.1002/wics.101.
- [Background] Cho YK, Lipowska AM, Nicodeme F, Teitelbaum EN, Hungness ES, Johnston ER, Gawron A, Kahrilas PJ, Pandolfino JE. Assessing bolus retention in achalasia using high-resolution manometry with impedance: a comparator study with timed barium esophagram. Am J Gastroenterol. 2014 Jun;109(6):829-35. doi: 10.1038/ajg.2014.61. Epub 2014 Apr 8. PMID 24710506
- [Background] Halland M, Ravi K, Barlow J, Arora A. Correlation between the radiological observation of isolated tertiary waves on an esophagram and findings on high-resolution esophageal manometry. Dis Esophagus. 2016 Jan;29(1):22-6. doi: 10.1111/dote.12292. Epub 2014 Oct 20. PMID 25327483
- [Background] Bedell A, Taft TH, Keefer L, Pandolfino J. Development of the Northwestern Esophageal Quality of Life Scale: A Hybrid Measure for Use Across Esophageal Conditions. Am J Gastroenterol. 2016 Apr;111(4):493-9. doi: 10.1038/ajg.2016.20. Epub 2016 Feb 16. PMID 26881974
- [Background] Cieslak MC, Castelfranco AM, Roncalli V, Lenz PH, Hartline DK. t-Distributed Stochastic Neighbor Embedding (t-SNE): A tool for eco-physiological transcriptomic analysis. Mar Genomics. 2020 Jun;51:100723. doi: 10.1016/j.margen.2019.100723. Epub 2019 Nov 26. PMID 31784353
- [Background] Acharya S, Kou W, Halder S, Carlson DA, Kahrilas PJ, Pandolfino JE, Patankar NA. Pumping Patterns and Work Done During Peristalsis in Finite-Length Elastic Tubes. J Biomech Eng. 2021 Jul 1;143(7):071001. doi: 10.1115/1.4050284. PMID 33625493
- [Background] Acharya S, Halder S, Carlson DA, Kou W, Kahrilas PJ, Pandolfino JE, Patankar NA. Assessment of esophageal body peristaltic work using functional lumen imaging probe panometry. Am J Physiol Gastrointest Liver Physiol. 2021 Feb 1;320(2):G217-G226. doi: 10.1152/ajpgi.00324.2020. Epub 2020 Nov 11. PMID 33174457
- [Background] Halder S, Acharya S, Kou W, Kahrilas PJ, Pandolfino JE, Patankar NA. Mechanics informed fluoroscopy of esophageal transport. Biomech Model Mechanobiol. 2021 Jun;20(3):925-940. doi: 10.1007/s10237-021-01420-0. Epub 2021 Mar 2. PMID 33651206
- [Background] Barnard AC, Hunt WA, Timlake WP, Varley E. A theory of fluid flow in compliant tubes. Biophys J. 1966 Nov;6(6):717-24. doi: 10.1016/S0006-3495(66)86690-0. PMID 5972373
- [Background] Holmstrom AL, Campagna RAJ, Cirera A, Carlson DA, Pandolfino JE, Teitelbaum EN, Hungness ES. Intraoperative use of FLIP is associated with clinical success following POEM for achalasia. Surg Endosc. 2021 Jun;35(6):3090-3096. doi: 10.1007/s00464-020-07739-6. Epub 2020 Jul 6. PMID 32632483
- [Background] Teitelbaum EN, Soper NJ, Pandolfino JE, Kahrilas PJ, Hirano I, Boris L, Nicodeme F, Lin Z, Hungness ES. Esophagogastric junction distensibility measurements during Heller myotomy and POEM for achalasia predict postoperative symptomatic outcomes. Surg Endosc. 2015 Mar;29(3):522-8. doi: 10.1007/s00464-014-3733-1. Epub 2014 Jul 24. PMID 25055891
- [Background] Yadlapati R, Hungness ES, Pandolfino JE. Complications of Antireflux Surgery. Am J Gastroenterol. 2018 Aug;113(8):1137-1147. doi: 10.1038/s41395-018-0115-7. Epub 2018 Jun 14. PMID 29899438
- [Background] Fibbe C, Layer P, Keller J, Strate U, Emmermann A, Zornig C. Esophageal motility in reflux disease before and after fundoplication: a prospective, randomized, clinical, and manometric study. Gastroenterology. 2001 Jul;121(1):5-14. doi: 10.1053/gast.2001.25486. PMID 11438489
- [Background] Paterson WG, Anderson MA, Anand N. Pharmacological characterization of lower esophageal sphincter relaxation induced by swallowing, vagal efferent nerve stimulation, and esophageal distention. Can J Physiol Pharmacol. 1992 Jul;70(7):1011-5. doi: 10.1139/y92-139. PMID 1360326
- [Background] Paterson WG. Esophageal and lower esophageal sphincter response to balloon distention in patients with achalasia. Dig Dis Sci. 1997 Jan;42(1):106-12. doi: 10.1023/a:1018893206926. PMID 9009124
- [Background] Carlson DA, Schauer JM, Kou W, Kahrilas PJ, Pandolfino JE. Functional Lumen Imaging Probe Panometry Helps Identify Clinically Relevant Esophagogastric Junction Outflow Obstruction per Chicago Classification v4.0. Am J Gastroenterol. 2023 Jan 1;118(1):77-86. doi: 10.14309/ajg.0000000000001980. Epub 2022 Aug 23. PMID 36002925
- [Background] Bredenoord AJ, Babaei A, Carlson D, Omari T, Akiyama J, Yadlapati R, Pandolfino JE, Richter J, Fass R. Esophagogastric junction outflow obstruction. Neurogastroenterol Motil. 2021 Sep;33(9):e14193. doi: 10.1111/nmo.14193. Epub 2021 Jun 12. PMID 34120375
- [Background] Agrawal A, Hila A, Tutuian R, Mainie I, Castell DO. Bethanechol improves smooth muscle function in patients with severe ineffective esophageal motility. J Clin Gastroenterol. 2007 Apr;41(4):366-70. doi: 10.1097/01.mcg.0000225542.03880.68. PMID 17413603
- [Background] Jandee S, Geeraerts A, Geysen H, Rommel N, Tack J, Vanuytsel T. Management of Ineffective Esophageal Hypomotility. Front Pharmacol. 2021 May 26;12:638915. doi: 10.3389/fphar.2021.638915. eCollection 2021. PMID 34122066
- [Background] Kessing BF, Smout AJ, Bennink RJ, Kraaijpoel N, Oors JM, Bredenoord AJ. Prucalopride decreases esophageal acid exposure and accelerates gastric emptying in healthy subjects. Neurogastroenterol Motil. 2014 Aug;26(8):1079-86. doi: 10.1111/nmo.12359. Epub 2014 May 29. PMID 24891067
- [Background] Camilleri M, Kerstens R, Rykx A, Vandeplassche L. A placebo-controlled trial of prucalopride for severe chronic constipation. N Engl J Med. 2008 May 29;358(22):2344-54. doi: 10.1056/NEJMoa0800670. PMID 18509121
- [Background] Lei WY, Hung JS, Liu TT, Yi CH, Chen CL. Influence of prucalopride on esophageal secondary peristalsis in reflux patients with ineffective motility. J Gastroenterol Hepatol. 2018 Mar;33(3):650-655. doi: 10.1111/jgh.13986. PMID 28898473
- [Background] Yi CH, Lei WY, Hung JS, Liu TT, Chen CL. Effects of prucalopride on esophageal secondary peristalsis in humans. Clin Transl Gastroenterol. 2016 Nov 10;7(11):e202. doi: 10.1038/ctg.2016.58. PMID 27831544
- [Background] Xiao Y, Kahrilas PJ, Nicodeme F, Lin Z, Roman S, Pandolfino JE. Lack of correlation between HRM metrics and symptoms during the manometric protocol. Am J Gastroenterol. 2014 Apr;109(4):521-6. doi: 10.1038/ajg.2014.13. Epub 2014 Feb 11. PMID 24513804
- [Background] Taft TH, Carlson DA, Simons M, Zavala S, Hirano I, Gonsalves N, Pandolfino JE. Esophageal Hypervigilance and Symptom-Specific Anxiety in Patients with Eosinophilic Esophagitis. Gastroenterology. 2021 Oct;161(4):1133-1144. doi: 10.1053/j.gastro.2021.06.023. Epub 2021 Jun 19. PMID 34153298
- [Background] Taft TH, Triggs JR, Carlson DA, Guadagnoli L, Tomasino KN, Keefer L, Pandolfino JE. Validation of the oesophageal hypervigilance and anxiety scale for chronic oesophageal disease. Aliment Pharmacol Ther. 2018 May;47(9):1270-1277. doi: 10.1111/apt.14605. Epub 2018 Mar 12. PMID 29528128
- [Background] Eckardt VF, Aignherr C, Bernhard G. Predictors of outcome in patients with achalasia treated by pneumatic dilation. Gastroenterology. 1992 Dec;103(6):1732-8. doi: 10.1016/0016-5085(92)91428-7. PMID 1451966
- [Background] Taft TH, Carlson DA, Triggs J, Craft J, Starkey K, Yadlapati R, Gregory D, Pandolfino JE. Evaluating the reliability and construct validity of the Eckardt symptom score as a measure of achalasia severity. Neurogastroenterol Motil. 2018 Jun;30(6):e13287. doi: 10.1111/nmo.13287. Epub 2018 Jan 8. PMID 29315993
- [Background] Taft TH, Riehl M, Sodikoff JB, Kahrilas PJ, Keefer L, Doerfler B, Pandolfino JE. Development and validation of the brief esophageal dysphagia questionnaire. Neurogastroenterol Motil. 2016 Dec;28(12):1854-1860. doi: 10.1111/nmo.12889. Epub 2016 Jul 5. PMID 27380834
- [Background] Halder S, Acharya S, Kou W, Campagna RAJ, Triggs JR, Carlson DA, Aadam AA, Hungness ES, Kahrilas PJ, Pandolfino JE, Patankar NA. Myotomy technique and esophageal contractility impact blown-out myotomy formation in achalasia: an in silico investigation. Am J Physiol Gastrointest Liver Physiol. 2022 May 1;322(5):G500-G512. doi: 10.1152/ajpgi.00281.2021. Epub 2022 Feb 16. PMID 35170365
- [Background] Triggs JR, Krause AJ, Carlson DA, Donnan EN, Campagna RAJ, Jain AS, Kahrilas PJ, Hungness ES, Pandolfino JE. Blown-out myotomy: an adverse event of laparoscopic Heller myotomy and peroral endoscopic myotomy for achalasia. Gastrointest Endosc. 2021 Apr;93(4):861-868.e1. doi: 10.1016/j.gie.2020.07.041. Epub 2020 Jul 25. PMID 32721488
- [Background] Nabi Z, Talukdar R, Mandavdhare H, Reddy DN. Short versus long esophageal myotomy during peroral endoscopic myotomy: A systematic review and meta-analysis of comparative trials. Saudi J Gastroenterol. 2022 Jul-Aug;28(4):261-267. doi: 10.4103/sjg.sjg_438_21. PMID 34806659
- [Background] Nabi Z, Ramchandani M, Sayyed M, Chavan R, Darisetty S, Goud R, Murthy HVV, Reddy DN. Comparison of Short Versus Long Esophageal Myotomy in Cases With Idiopathic Achalasia: A Randomized Controlled Trial. J Neurogastroenterol Motil. 2021 Jan 30;27(1):63-70. doi: 10.5056/jnm20022. PMID 32675389
- [Background] Sifrim D, Janssens J. Secondary peristaltic contractions, like primary peristalsis, are preceded by inhibition in the human esophageal body. Digestion. 1996;57(1):73-8. doi: 10.1159/000201316. PMID 8626052
- [Background] Halder S, Pandolfino JE, Kahrilas PJ, Koop A, Schauer J, Araujo IK, Elisha G, Kou W, Patankar NA, Carlson DA. Assessing mechanical function of peristalsis with functional lumen imaging probe panometry: Contraction power and displaced volume. Neurogastroenterol Motil. 2023 Dec;35(12):e14692. doi: 10.1111/nmo.14692. Epub 2023 Oct 16. PMID 37845833
- [Background] Acharya S, Halder S, Carlson DA, Kou W, Kahrilas PJ, Pandolfino JE, Patankar NA. Estimation of mechanical work done to open the esophagogastric junction using functional lumen imaging probe panometry. Am J Physiol Gastrointest Liver Physiol. 2021 May 1;320(5):G780-G790. doi: 10.1152/ajpgi.00032.2021. Epub 2021 Mar 3. PMID 33655760
- [Background] Kou W, Carlson DA, Patankar NA, Kahrilas PJ, Pandolfino JE. Four-dimensional impedance manometry derived from esophageal high-resolution impedance-manometry studies: a novel analysis paradigm. Therap Adv Gastroenterol. 2020 Oct 24;13:1756284820969050. doi: 10.1177/1756284820969050. eCollection 2020. PMID 33178334
- [Background] Carlson DA, Kahrilas PJ, Lin Z, Hirano I, Gonsalves N, Listernick Z, Ritter K, Tye M, Ponds FA, Wong I, Pandolfino JE. Evaluation of Esophageal Motility Utilizing the Functional Lumen Imaging Probe. Am J Gastroenterol. 2016 Dec;111(12):1726-1735. doi: 10.1038/ajg.2016.454. Epub 2016 Oct 11. PMID 27725650
- [Background] Vespa E, Farina DA, Kahrilas PJ, Kou W, Low EE, Yadlapati R, Pandolfino JE, Carlson DA. Identifying spastic variant of type II achalasia after treatment with high-resolution manometry and FLIP Panometry. Neurogastroenterol Motil. 2023 Jul;35(7):e14552. doi: 10.1111/nmo.14552. Epub 2023 Feb 21. PMID 36807659
- [Background] Low EE, Fehmi SA, Hasan A, Chang M, Kwong W, Krinsky ML, Anand G, Greytak M, Kaizer A, Carlson DA, Pandolfino JE, Yadlapati R. Type II achalasia with focal elevated pressures: A distinct manometric and clinical sub-group. Neurogastroenterol Motil. 2022 Dec;34(12):e14449. doi: 10.1111/nmo.14449. Epub 2022 Aug 16. PMID 35972282
- [Background] Rohof WO, Salvador R, Annese V, Bruley des Varannes S, Chaussade S, Costantini M, Elizalde JI, Gaudric M, Smout AJ, Tack J, Busch OR, Zaninotto G, Boeckxstaens GE. Outcomes of treatment for achalasia depend on manometric subtype. Gastroenterology. 2013 Apr;144(4):718-25; quiz e13-4. doi: 10.1053/j.gastro.2012.12.027. Epub 2012 Dec 28. PMID 23277105
- [Background] Pandolfino JE, Kwiatek MA, Nealis T, Bulsiewicz W, Post J, Kahrilas PJ. Achalasia: a new clinically relevant classification by high-resolution manometry. Gastroenterology. 2008 Nov;135(5):1526-33. doi: 10.1053/j.gastro.2008.07.022. Epub 2008 Jul 22. PMID 18722376
- [Background] Richardson C, Agrawal R, Lee J, Almagor O, Nelson R, Varga J, Cuttica MJ, Dematte JD, Chang RW, Hinchcliff ME. Esophageal dilatation and interstitial lung disease in systemic sclerosis: A cross-sectional study. Semin Arthritis Rheum. 2016 Aug;46(1):109-14. doi: 10.1016/j.semarthrit.2016.02.004. Epub 2016 Feb 26. PMID 27033049
- [Background] Jain AS, Carlson DA, Triggs J, Tye M, Kou W, Campagna R, Hungness E, Kim D, Kahrilas PJ, Pandolfino JE. Esophagogastric Junction Distensibility on Functional Lumen Imaging Probe Topography Predicts Treatment Response in Achalasia-Anatomy Matters! Am J Gastroenterol. 2019 Sep;114(9):1455-1463. doi: 10.14309/ajg.0000000000000137. PMID 30741739
- [Background] Carlson DA, Prescott JE, Germond E, Brenner D, Carns M, Correia CS, Tetreault MP, McMahan ZH, Hinchcliff M, Kou W, Kahrilas PJ, Perlman HR, Pandolfino JE. Heterogeneity of primary and secondary peristalsis in systemic sclerosis: A new model of "scleroderma esophagus". Neurogastroenterol Motil. 2022 Jul;34(7):e14284. doi: 10.1111/nmo.14284. Epub 2021 Oct 28. PMID 34709690
- [Background] Carlson DA, Gyawali CP, Khan A, Yadlapati R, Chen J, Chokshi RV, Clarke JO, Garza JM, Jain AS, Katz P, Konda V, Lynch K, Schnoll-Sussman FH, Spechler SJ, Vela MF, Prescott JE, Baumann AJ, Donnan EN, Kou W, Kahrilas PJ, Pandolfino JE. Classifying Esophageal Motility by FLIP Panometry: A Study of 722 Subjects With Manometry. Am J Gastroenterol. 2021 Dec 1;116(12):2357-2366. doi: 10.14309/ajg.0000000000001532. PMID 34668487
- [Background] Carlson DA, Kou W, Lin Z, Hinchcliff M, Thakrar A, Falmagne S, Prescott J, Dorian E, Kahrilas PJ, Pandolfino JE. Normal Values of Esophageal Distensibility and Distension-Induced Contractility Measured by Functional Luminal Imaging Probe Panometry. Clin Gastroenterol Hepatol. 2019 Mar;17(4):674-681.e1. doi: 10.1016/j.cgh.2018.07.042. Epub 2018 Aug 3. PMID 30081222
- [Background] Nguyen AD, Ellison A, Reddy CA, Mendoza R, Podgaetz E, Ward MA, Souza RF, Spechler SJ, Konda VJA. Spastic secondary contractile patterns identified by FLIP panometry in symptomatic patients with unremarkable high-resolution manometry. Neurogastroenterol Motil. 2022 Jul;34(7):e14321. doi: 10.1111/nmo.14321. Epub 2022 Jan 24. PMID 35075734
- [Background] Omari TI, Zifan A, Cock C, Mittal RK. Distension contraction plots of pharyngeal/esophageal peristalsis: next frontier in the assessment of esophageal motor function. Am J Physiol Gastrointest Liver Physiol. 2022 Sep 1;323(3):G145-G156. doi: 10.1152/ajpgi.00124.2022. Epub 2022 Jul 5. PMID 35788152
- [Background] Choi JY, Jung KW, Pandolfino JE, Choi K, Park YS, Na HK, Ahn JY, Lee JH, Kim DH, Choi KD, Song HJ, Lee GH, Jung HY. Dysphagia associated with esophageal wall thickening in patients with nonspecific high-resolution manometry findings: Understanding motility beyond the Chicago classification version 4.0. Neurogastroenterol Motil. 2024 Apr;36(4):e14736. doi: 10.1111/nmo.14736. Epub 2024 Jan 15. PMID 38225864
- [Background] Carlson DA, Lin Z, Rogers MC, Lin CY, Kahrilas PJ, Pandolfino JE. Utilizing functional lumen imaging probe topography to evaluate esophageal contractility during volumetric distention: a pilot study. Neurogastroenterol Motil. 2015 Jul;27(7):981-9. doi: 10.1111/nmo.12572. Epub 2015 Apr 20. PMID 25898916
- [Background] Lin Z, Yim B, Gawron A, Imam H, Kahrilas PJ, Pandolfino JE. The four phases of esophageal bolus transit defined by high-resolution impedance manometry and fluoroscopy. Am J Physiol Gastrointest Liver Physiol. 2014 Aug 15;307(4):G437-44. doi: 10.1152/ajpgi.00148.2014. Epub 2014 Jun 26. PMID 24970774
- [Background] Kou W, Carlson DA, Kahrilas PJ, Patankar NA, Pandolfino JE. Normative values of intra-bolus pressure and esophageal compliance based on 4D high-resolution impedance manometry. Neurogastroenterol Motil. 2022 Oct;34(10):e14423. doi: 10.1111/nmo.14423. Epub 2022 Jun 5. PMID 35661346
- [Background] Aziz Q, Fass R, Gyawali CP, Miwa H, Pandolfino JE, Zerbib F. Functional Esophageal Disorders. Gastroenterology. 2016 Feb 15:S0016-5085(16)00178-5. doi: 10.1053/j.gastro.2016.02.012. Online ahead of print. PMID 27144625
- [Background] Carlson DA, Gyawali CP, Roman S, Vela M, Taft TH, Crowell MD, Ravi K, Triggs JR, Quader F, Prescott J, Lin FTJ, Mion F, Biasutto D, Keefer L, Kahrilas PJ, Pandolfino JE. Esophageal Hypervigilance and Visceral Anxiety Are Contributors to Symptom Severity Among Patients Evaluated With High-Resolution Esophageal Manometry. Am J Gastroenterol. 2020 Mar;115(3):367-375. doi: 10.14309/ajg.0000000000000536. PMID 31990697
- [Background] Monrroy H, Cisternas D, Bilder C, Ditaranto A, Remes-Troche J, Meixueiro A, Zavala MA, Serra J, Marin I, Ruiz de Leon A, Perez de la Serna J, Hani A, Leguizamo A, Abrahao L, Coello R, Valdovinos MA. The Chicago Classification 3.0 Results in More Normal Findings and Fewer Hypotensive Findings With No Difference in Other Diagnoses. Am J Gastroenterol. 2017 Apr;112(4):606-612. doi: 10.1038/ajg.2017.10. Epub 2017 Jan 31. PMID 28139656
- [Background] Clouse RE, Staiano A. Topography of the esophageal peristaltic pressure wave. Am J Physiol. 1991 Oct;261(4 Pt 1):G677-84. doi: 10.1152/ajpgi.1991.261.4.G677. PMID 1928353
- [Background] Halder S, Yamasaki J, Acharya S, Kou W, Elisha G, Carlson DA, Kahrilas PJ, Pandolfino JE, Patankar NA. Virtual disease landscape using mechanics-informed machine learning: Application to esophageal disorders. Artif Intell Med. 2022 Dec;134:102435. doi: 10.1016/j.artmed.2022.102435. Epub 2022 Oct 31. PMID 36462900
- [Background] Koop AH, Kahrilas PJ, Schauer J, Pandolfino JE, Carlson DA. The impact of primary peristalsis, contractile reserve, and secondary peristalsis on esophageal clearance measured by timed barium esophagogram. Neurogastroenterol Motil. 2023 Oct;35(10):e14638. doi: 10.1111/nmo.14638. Epub 2023 Jul 7. PMID 37417394
- [Background] Carlson DA, Baumann AJ, Donnan EN, Krause A, Kou W, Pandolfino JE. Evaluating esophageal motility beyond primary peristalsis: Assessing esophagogastric junction opening mechanics and secondary peristalsis in patients with normal manometry. Neurogastroenterol Motil. 2021 Oct;33(10):e14116. doi: 10.1111/nmo.14116. Epub 2021 Mar 11. PMID 33705590
- [Background] Carlson DA, Kou W, Masihi M, Acharya S, Baumann AJ, Donnan EN, Kahrilas PJ, Pandolfino JE. Repetitive Antegrade Contractions: A novel response to sustained esophageal distension is modulated by cholinergic influence. Am J Physiol Gastrointest Liver Physiol. 2020 Oct 7. doi: 10.1152/ajpgi.00305.2020. Online ahead of print. PMID 33026823
- [Background] Carlson DA, Kathpalia P, Craft J, Tye M, Lin Z, Kahrilas PJ, Pandolfino JE. The relationship between esophageal acid exposure and the esophageal response to volumetric distention. Neurogastroenterol Motil. 2018 Mar;30(3):10.1111/nmo.13240. doi: 10.1111/nmo.13240. Epub 2017 Nov 2. PMID 29098750
- [Background] Carlson DA, Lin Z, Kahrilas PJ, Sternbach J, Donnan EN, Friesen L, Listernick Z, Mogni B, Pandolfino JE. The Functional Lumen Imaging Probe Detects Esophageal Contractility Not Observed With Manometry in Patients With Achalasia. Gastroenterology. 2015 Dec;149(7):1742-51. doi: 10.1053/j.gastro.2015.08.005. Epub 2015 Aug 14. PMID 26278501
- [Background] Yadlapati R, Kahrilas PJ, Fox MR, Bredenoord AJ, Prakash Gyawali C, Roman S, Babaei A, Mittal RK, Rommel N, Savarino E, Sifrim D, Smout A, Vaezi MF, Zerbib F, Akiyama J, Bhatia S, Bor S, Carlson DA, Chen JW, Cisternas D, Cock C, Coss-Adame E, de Bortoli N, Defilippi C, Fass R, Ghoshal UC, Gonlachanvit S, Hani A, Hebbard GS, Wook Jung K, Katz P, Katzka DA, Khan A, Kohn GP, Lazarescu A, Lengliner J, Mittal SK, Omari T, Park MI, Penagini R, Pohl D, Richter JE, Serra J, Sweis R, Tack J, Tatum RP, Tutuian R, Vela MF, Wong RK, Wu JC, Xiao Y, Pandolfino JE. Esophageal motility disorders on high-resolution manometry: Chicago classification version 4.0(c). Neurogastroenterol Motil. 2021 Jan;33(1):e14058. doi: 10.1111/nmo.14058. PMID 33373111
- [Background] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Background] Pandolfino JE, Ghosh SK, Rice J, Clarke JO, Kwiatek MA, Kahrilas PJ. Classifying esophageal motility by pressure topography characteristics: a study of 400 patients and 75 controls. Am J Gastroenterol. 2008 Jan;103(1):27-37. doi: 10.1111/j.1572-0241.2007.01532.x. Epub 2007 Sep 26. PMID 17900331
- [Background] Peery AF, Crockett SD, Murphy CC, Jensen ET, Kim HP, Egberg MD, Lund JL, Moon AM, Pate V, Barnes EL, Schlusser CL, Baron TH, Shaheen NJ, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2021. Gastroenterology. 2022 Feb;162(2):621-644. doi: 10.1053/j.gastro.2021.10.017. Epub 2021 Oct 19. PMID 34678215